CLINICAL TRIAL: NCT02792088
Title: A Phase III, Multi-center, Randomized, Double-blinded, Parallel Study to Assess the Antiviral Activity and Safety Endpoints for the Treatment of Besifovir 150mg Compared to Tenofovir 300mg in Chronic Hepatitis B Patients Who Have Resistance to Nucleoside Analogues
Brief Title: Study to Assess the Antiviral Activity and Safety Endpoints for the Treatment of Besifovir 150mg Compared to Tenofovir 300mg in Chronic Hepatitis B Patients Who Have Resistance to Nucleoside Analogues
Acronym: HBV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID_BVCL012
Record Dates: First submitted 2016-05-31; First posted 2016-06-07 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis B
Keywords: HBV
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — ((1-((2-amino-9H-purin-9-yl)methyl)cyclopropyl)oxy)methylphosphonic acid dipivoxyl; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Besifovir (Experimental): Besifovir 150 mg q.d.
  Interventions: Drug: Besifovir 150mg
- Tenofovir (Active Comparator): Tenofovir 300 mg q.d.
  Interventions: Drug: Tenofovir 300mg

INTERVENTIONS:
Drug: Besifovir 150mg — Besifovir 150 mg q.d. + Placebo of Tenofovir Disoproxil Fumarate 300 mg q.d. + L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Other Names: Besifovir
  Arms: Besifovir
Drug: Tenofovir 300mg — Placebo of Besifovir 150 mg q.d. + Tenofovir Disoproxil Fumarate 300 mg q.d. + Placebo of L-carnitine (L-Carn Tab. 330 mg) 660 mg q.d.
  Other Names: Tenofovir
  Arms: Tenofovir

SUMMARY:
To prove that a study drug is noninferior to a control drug with a proportion of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) at the 48th week after 48-week administration of Besifovir 150 mg, or Tenofovir 300 mg as a control drug to chronic hepatitis B patients

DETAILED DESCRIPTION:
* Screening Period Subject registration is conducted with confirming selection and exclusion criteria after a written consent form is obtained within 42 days before clinical trial drug administration.
* Baseline Subjects who visit on the date of starting clinical trial drug administration are randomized to a test group or a control group at a ratio of 1:1. Double blindness is applied for both groups.
* Treatment period Subjects are orally administered with a clinical trial drug q.ds.i.d. for 48 weeks and visit at the 0, 4th, 12th, 24th, 36th, and 48th week for an HBV DNA test, laboratory tests, a physical test, vital signs, and adverse events.
* Follow-up period Subjects are provided with appropriate treatment after completing the 48-week trial or dropping out. Subjects visit once at the 60th week for follow-up of adverse events, such as acute deterioration of hepatitis B, and HBV DNA test results. If any treatment is not conducted after 48-week administration, subjects visit at intervals of four weeks until a follow-up visit (60th week) and the same tests with the 24th week visit (Visit 5) are conducted. However, subjects who participate in a 48-week separate extended trial conducted after 48-week administration in this clinical trial do not have a follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who show positive HBsAg or has a history of chronic hepatitis B for the last six months or more before screening
* Patients who showed positive HBsAg during screening
* Have developed nucleoside analogue resistant HB
* Had no received nucleotide analogue

Exclusion Criteria:

1. Treatment with pegylated interferons within 6 months
2. Prior exposure to BSV
3. Mutations conferring resistance to ADV
4. Serum HBV DNA levels < 69 IU/mL
5. Coinfection with hepatitis C, hepatitis D or human immunodeficiency viruses
6. ALT levels ≥ 10 x ULN
7. Evidence of decompensated liver disease (Total bilirubin > 2 x ULN, prothrombin time > 6 sec prolonged or INR >1.5, serum albumin <2.8 g/dL, uncontrolled ascites, overt hepatic encephalopathy, or Child-Pugh score ≥8)
8. Certain laboratory abnormalities (Hemoglobin < 9.0 g/dL, absolute neutrophil count (ANC) < 1 x 109/L (1000/mm3), platelet count < 75 x 109/L (75 x 103/mm3), serum Creatinine > 1.5 mg/dL, or serum amylase > 2 x ULN and Lipase > 2 x ULN)
9. Decreased estimated glomerular filtration rates < 50 mL/min
10. Presence of hepatocellular carcinoma or elevated alpha feto-protein > 50 ng/mL
11. Current use of aspirin or nonsteroidal anti-inflammatory drugs within 2 month
12. Current use of immunosuppressive agents within 6 months
13. Current use of high dose corticosteroids (prednisolone > 20 mg/day or equivalent dose over 14 days) with 3 months
14. History of malignancy within 5 years
15. Subjects who are participating in other clinical trials
16. Pregnant or lactating women
17. Hypersensitivity to the study drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
The rate of subjects who showed HBV DNA undetected (less than 400 copies/mL (69 IU/mL)) at the 48th week | at the 48th week

SECONDARY OUTCOMES:
The rate of subjects who showed ALT normalized at the 48th week | at the 48th week

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Hyub Han, M.D, Ph.D., Principal Investigator — Severance Hospital of Yonsei University
Locations (1):
- Severance Hospital of Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided